CLINICAL TRIAL: NCT02620033
Title: Impact of Yoga As Complementary Therapy on Quality of Life, Pro-inflammatory, and Cellular Immune Biomarkers in Patients Undergoing Radical Prostatectomy: A Pilot Randomized-Controlled Trial
Brief Title: Impact of Yoga As Complementary Therapy in Patients Undergoing Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC2015-406H
Record Dates: First submitted 2015-10-15; First posted 2015-12-02 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy; Yoga therapy; Health related quality of life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Those assigned to the standard care group will follow the routine pre- and post-operative care for patients whose undergoing radical prostatectomy.
- Yoga therapy group (Active Comparator): Those assigned to the yoga therapy group will be asked to participate in yoga session three times in a week for 6 weeks prior to the scheduled surgery and then re-initiated 3 weeks after the surgery for another 6 weeks. Each session will be approximately 60 - 75 minutes. These yoga session will be held at Nydia's Yoga Therapy Studio, located in San Antonio, TX, under the guidance of certified yoga instructor, Dr. Nydia Tijerina Darby, PT, DPT, MS, who's the owner of the studio and co-investigator of this study. The yoga exercise will be tailored to patient's comfort level.
  Interventions: Behavioral: Yoga therapy

INTERVENTIONS:
Behavioral: Yoga therapy
  Arms: Yoga therapy group

SUMMARY:
The researchers hope to learn if yoga complementary therapy would improve health-related quality of life, recovery of urinary continence and erectile function in patients who underwent prostate cancer surgery (i.e. radical prostatectomy). We hypothesized that in patients undergoing radical prostatectomy, preoperative and postoperative Yoga complementary therapy would improve health- related quality of life (HRQOL), recovery of urinary continence and erectile function.

This two-arm, randomized controlled pilot study will compare Yoga intervention to usual care group. The aim is to evaluate the efficacy of Yoga complementary therapy on HRQOL in patients who underwent radical prostatectomy (RP). Yoga therapy will be given to the intervention group three times in a week for 6 weeks prior to surgery and then initiated 3 weeks after the surgery for another 6 weeks. The yoga exercise will be tailored to the participant's comfort level. As an exploratory analysis, we will evaluate pro-inflammatory and immunological markers.

ELIGIBILITY:
Inclusion Criteria:

* Men between the age of 30 to 80
* Has been diagnosed with localized prostate cancer (i.e. pathologically and/or radiographically confirmed)
* Is scheduled to undergo radical prostatectomy (i.e. robot-assisted or open-approach)
* Has no other active primary malignancy aside from prostate cancer
* Currently not practicing yoga as a form of exercise and/or meditation
* Does not have uncontrolled pain
* Does not have neurological or musculoskeletal co-morbidity inhibiting exercise
* Has never been diagnosed by health care professionals to have absolute contraindications to exercise testing
* Willing to be randomized to either standard care or intervention group
* Willing to participate in yoga therapy for twelve weeks if randomized to intervention group
* Willing to undergo phlebotomy
* Able and willing to provide informed consent

Exclusion Criteria:

* Men under the age of 30 or over the age of 80
* Has NOT been diagnosed with localized prostate cancer (i.e. pathologically and/or radiographically confirmed)
* Is NOT scheduled to undergo radical prostatectomy (i.e. robot-assisted or open-approach)
* Has other active primary malignancy aside from prostate cancer
* Currently practicing yoga as a form of exercise and/or meditation
* Has uncontrolled pain
* Has neurological or musculoskeletal co-morbidity inhibiting exercise
* Has been diagnosed with psychotic, addictive, and major cognitive disorders
* Has been diagnosed by health care professionals to have absolute contraindications to exercise testing Unwilling to be randomized to either standard care or intervention group
* Unwilling to participate in yoga therapy for twelve weeks if randomized to intervention group
* Unwilling to undergo phlebotomy
* Unable and unwilling to provide informed consent

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health related quality of life measures | One year
  health related quality of life measures including but not limited to fatigue level, recovery urinary continence, and erectile function.
Change from baseline in 6-minute walk test | One year
Total number of participants recruited to and withdraw from the study | One year
Total number of participants completed the study | One year
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | One year

SECONDARY OUTCOMES:
Change from baseline level on pro-inflammatory biomarkers | one year
Change from baseline level on cellular immune response (i.e. measuring the Natural Killer Cell and regulatory-T cells) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Dharam Kaushik, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Result] Kaushik D, Shah PK, Mukherjee N, Ji N, Dursun F, Kumar AP, Thompson IM Jr, Mansour AM, Jha R, Yang X, Wang H, Darby N, Ricardo Rivero J, Svatek RS, Liss MA. Effects of yoga in men with prostate cancer on quality of life and immune response: a pilot randomized controlled trial. Prostate Cancer Prostatic Dis. 2022 Sep;25(3):531-538. doi: 10.1038/s41391-021-00470-w. Epub 2021 Nov 23. PMID 34815548